CLINICAL TRIAL: NCT03309891
Title: A Phase 2, Randomized, Open-label, Active Controlled, Dose Finding Study of Long-acting Hybrid Fc Fused Recombinant Human Growth Hormone (GX-H9) in Paeditaric Patients With Growth Hormone Deficiency
Brief Title: Dose Finding Study of GX-H9 in Paeditaric Patients With Growth Hormone Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX-H9-003
Record Dates: First submitted 2017-09-05; First posted 2017-10-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — GX-H9; Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: A Phase 2, randomized, open-label, active controlled, dose finding study
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): GX-H9 subcutaneous injections (weekly)
  Interventions: Drug: GX-H9
- Cohort 2 (Experimental): GX-H9 subcutaneous injections (weekly)
  Interventions: Drug: GX-H9
- Cohort 3 (Experimental): GX-H9 subcutaneous injections (twice-monthly)
  Interventions: Drug: GX-H9
- Cohort 4 (Active Comparator): Genotropin subcutaneous injections (daily)
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: GX-H9 — subcutaneous injection (weekly or twice-monthly)
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Genotropin — subcutaneous injection (daily)
  Arms: Cohort 4

SUMMARY:
This is a randomized, open-label, active controlled, Phase 2 study designed to assess the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of weekly and semi-monthly doses of GX-H9 in the treatment of Paediatric Growth Hormone Deficiency (PGHD) as compared to the standard of care daily rhGH treatment.

DETAILED DESCRIPTION:
GX-H9 is a new hGH product fused to hybrid Fc in studies as a once-a-week and every other week dosing regimen designed to overcome the inconvenience of daily rhGH injections and is under the studies designed to determine if the safety profile is comparable to currently approved daily rhGH products. Obviating the need for daily injections may increase compliance and therefore efficacy, which would be of great benefit to both paediatric and adult patients with GHD and other disorders with associated growth impairment and need for hGH substitution.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-pubertal children with either isolated GHD, or GH insufficiency as part of multiple pituitary hormone insufficiency, idiopathic or organic GH insufficiency (e.g., due to pituitary tumor, pituitary or brain surgery):

   * Boys: 3 years ≤ boy's age ≤ 11 years
   * Girls: 3 years ≤ girl's age ≤ 10 years
2. GHD confirmed by 2 different GH provocation tests with peak GH concentration below 10 ng/mL as described in consensus guidelines. Well documented historical GH provocation tests can be used for study eligibility providing that the tests are performed as defined in Appendix 2 (e.g. the same sampling time points). Data of each historical GH stimulation test will be reviewed by Medical Monitor and Sponsor in order to assess acceptance for the study
3. Without prior exposure to any rhGH therapy
4. Bone age (BA) is not older than chronological age and should not be greater than 9 years for girls and 10 years for boys
5. Impaired height and height velocity defined as:

   * Height (HT) of at least 2.0 standard deviations (SD) below the mean height for chronological age (CA) and gender according to the standards from Prader et. al 1989, (HT SDS ≤ -2.0)
   * Annualized height velocity (HV) of at least 1 SD below the mean HV for chronological age and gender according to the standards of Prader et al (1989). The interval between two height measurements should be at least 6 months (but not longer than 18 months) before inclusion
6. All subjects must have at least one cranial imaging study [magnetic resonance imaging (MRI) or computed tomography (CT)] prior to randomization:

   * To exclude intracranial causes of GHD in subjects without history of pituitary tumor [obtained within 6 months prior to informed consent signing, or
   * Subjects with a previously treated pituitary tumor must have no tumor progression for at least the past year [obtained within 3 months prior to informed consent signing, compared with a previous MRI or CT performed at least 12 months earlier]
   * If not performed within these specified time frames prior to informed consent signing, may be performed as a part of the screening procedures
7. Body mass Index (BMI) must be within ±2 SD of mean BMI for the chronological age and sex according to the 2000 CDC standards
8. Baseline IGF-1 level of at least 1 SD below the mean IGF-1 level standardized for age and sex (IGF-1 SDS≤ -1.0) according to the central laboratory reference values. One IGF-1 retest is allowed during the Screening period if first results were not higher than

   -0.85 SDS and if GH stimulation tests results and auxology parameters met eligibility criteria
9. Children with normal fundoscopy (ophthalmoscopy) at screening (without signs/symptoms of intracranial hypertension as assessed by fundoscopy) - it is highly recommended to take a photograph (if equipment is available at the study center)
10. Children with multiple hormonal deficiencies must be on stable replacement therapies for other hypothalamo-pituitary-organ axes for at least 3 months and 6 months for thyroid replacement therapy prior to Screening. Temporary adjustment of glucocorticoid replacement therapy, as appropriate, is acceptable
11. Normal 46 XX karyotype for girls
12. Written informed consent of the parent or legal guardian of the subject and assent of the subject (if the subject can read)
13. Parent or legal guardian who is capable and willing to administer the study drug

Exclusion Criteria:

1. History of radiation therapy or chemotherapy
2. Malnourished children defined as:

   * Serum albumin below the lower limit of normal (LLN) according to the reference ranges of central laboratory; and
   * Serum iron below the lower limit of normal (LLN) according to the reference ranges of central laboratory; and
   * BMI<-2 SD for age and sex
3. Children with psychosocial dwarfism
4. Children born small for gestational age (SGA-birth weight and/or birth length < -2 SD for gestational age according to the standards from Niklasson et al., 1991)
5. Presence of anti-hGH antibodies at screening
6. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, etc.
7. Subjects with diabetes mellitus
8. Subjects with impaired fasting sugar (based on WHO; fasting blood sugar > 110mg/dl or 6.1 mmol/l) after repeated blood analysis
9. Chromosomal abnormalities and medical syndromes (Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, SHOX mutations/deletions and skeletal dysplasias), with the exception of septo-optic dysplasia
10. Evidence of closed epiphyses
11. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids and methylphenidate for attention deficit hyperactivity disorder (ADHD), with the exception of hormone replacement therapies [thyroxine, hydrocortisone, desmopressin (DDAVP)]
12. Children requiring glucocorticoid therapy, other than treated for hypothalamo-pituitary-adrenal insufficiency in replacement doses who are taking a dose of greater than 400 μg/d of inhaled budesonide or equivalents for longer than 1 month during a calendar year (e.g. asthma)
13. Major medical conditions and/or presence of contraindication to rhGH treatment
14. Has a history of positive serology results to HIV, HBV and/or HCV
15. Subject who has a known or suspected hypersensitivity to rhGH
16. Other causes of short stature such as coeliac disease, hypothyroidism and rickets
17. The subject and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct
18. Subject who has received an investigational product, or has participated in a clinical study within 60 days before screening

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Annual height velocity in cm/year | 6 months
  The primary efficacy variable was the AHV in cm/year at 6 months.

SECONDARY OUTCOMES:
Annualized Height velocity expressed in SDS | 3, 6, 12 and 24 months
Change in height SDS (compared to baseline value) | 3, 6, 12 and 24 months
Annualized height velocity expressed in cm/year | 3, 12 and 24 months
Change in height expressed in cm | 3, 6, 12 and 24 months
Change in absolute IGF-I levels | 25 months
Change in IGF-I SDS | 25 months
Change in absolute IGFBP-3 levels | 25 months
Change in IGFBP-3 SDS | 25 months
Bone maturation after 12 and 24 months of treatment; | 12 and 24 months
Predicted adult height change from start to 12 and 24 months | 12 and 24 months
Number of subjects needing at least one dose modification | 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Jungwon Woo, Study Director — Genexine, Inc.
Locations (1):
- Odessa National Medical University, Odessa Regional Children's Hospital, Odesa, Ukraine